CLINICAL TRIAL: NCT04016636
Title: "Impact of Ibrutinib on the Quality of Life (QOL) in Patients With Chronic Lymphocytic Leukemia (CLL): Argentinian Experience"
Brief Title: A Study to Evaluate Impact of Ibrutinib on the Quality of Life (QOL) in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Mela Osorio Maria Jose (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Mela Osorio Maria Jose, Principal Investigator, Fundaleu
Organization: Fundaleu (Other)
Other Study IDs: QOL-Fundaleu0819
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: CLL
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Study. Patients with CLL receiving ibrutinib.: In this study the investigator does not assign specific interventions to the study participants. Participants will receive interventions as part of routine medical care, and the investigator will observe the effect of the intervention.
  This study will collect prospective real-world data to describe the quality of life (QOL) in patients with CLL receiving ibrutinib in routine Argentinian clinical practice over a 12-month follow-up period.
  The primary data source for this observational study will be the medical records of each enrolled patient, as well as questionnaires concerning quality of life. Data will be collected at baseline and on months 1,3,6 and 12 during a prospective period.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Participants in this observational study with confirmed diagnosis of CLL receiving ibrutinib in routine clinical practice settings will be observed approximately for 12 months.

SUMMARY:
The aim of this study is to evaluate the impact of Ibrutinib monotherapy in the QoL of subjects with Chronic Lymphocytic Leukemia (CLL) based in European Quality of Life 5 Dimensions (EQ-5D) and FACIT- fatigue questionnaires assessment from baseline to 1 year of treatment in Argentinian routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to any screening procedure
* Patients 18 years or older, to be treated with Ibrutinib, able to answer the complete QoL questionnaires.
* Diagnosis of CLL, according to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria, with pathology confirmation (World Health Organization 2008).
* Patients with CLL in first-line or with prior therapies or treatment-naïve patients that harbours deletion 17p according to fluorescence in situ hybridization (FISH) standards with an indication of treatment with ibrutinib.

Exclusion Criteria:

* Pregnant and breast-feeding patients
* Impairment of ingestion and/or absorption of ibrutinib
* Mental or physical limitation to complete the QoL questionnaires.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study includes patients with diagnosis of CLL with prescribed ibrutinib monotherapy as first-line or with prior therapies before or on the enrollment day as per routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Change From Baseline | 6 months
  The FACIT (Functional Assessment of Chronic Illness Therapy) fatigue scale is a self-assessment questionnaire with a 7-day recall period and 13 items evaluating fatigue and its impact on daily life activities. Fatigue is scored 0-52. 0= severe fatigue; 52= no fatigue.
  Number of patients with an improvement of at least 3 points in FACIT score (Minimally Important Difference).
  This study is assessing a Change from Baseline Fatigue at 6 months.

SECONDARY OUTCOMES:
Health-Related Quality of Life as Measured by European Quality of Life-5 Dimensions; 5 Levels Questionnaire (EQ-5D-5L) | At 0,1,3,6,12 months
  The EQ-5D questionnaire is a brief, generic health-related quality of life assessment (HRQOL) that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health).
  Number of patients with improvements in the EQ5D domains by analyzing the variation in each domain and index during follow-up at different time points.

OTHER OUTCOMES:
Number of patients with Clinically Significant Change in hemoglobin | At 0,1,3,6,12 months
  Number of Participants with Clinically Significant Change in hemoglobin will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jose Mela, MD, Principal Investigator — Fundaleu; Miguel A Pavlovsky, MD, Study Director — Fundaleu
Locations (1):
- Fundaleu, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided